CLINICAL TRIAL: NCT00472355
Title: Does Presynaptic Dopamine Receptor Stimulation Transiently Worsen Parkinsonism?
Brief Title: Low Dose Apomorphine and Parkinsonism
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient study materials
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, John G. Nutt, Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS021062 (NIH); M01RR000334 (NIH)
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; PD; apomorphine
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

INTERVENTIONS:
Drug: apomorphine

SUMMARY:
The purpose of this study is to determine if low doses of apomorphine worsen the motor symptoms of Parkinson's disease.

DETAILED DESCRIPTION:
The goal of the study is to learn why some people with Parkinson's disease (PD) get worse right after taking PD medication such as carbidopa/levodopa or as the medication is wearing off.

In this study scientists will determine if apomorphine, a drug used to treat symptoms of PD, will worsen the motor symptoms of people with PD when low doses of the drug are given as a continuous subcutaneous infusion. A continuous subcutaneous infusion means the drug is administered continuously through a small needle placed under the skin. Apomorphine, a PD drug that works similar to carbidopa/levodopa, will be used in this study because it is faster-acting and has a more brief effect than carbidopa/levodopa.

After the initial screening, participants will enter a 3-day treatment phase during which they will receive in random order low dose apomorphine, high dose apomorphine, or placebo (inactive substance). All participants will receive the study drug for 2 of the days at 2 different doses (low and high) and a placebo for 1 day. During the 3 days participants will provide blood samples and have their hearts monitored. Parkinsonism will be monitored each day by speed of finger tapping, foot tapping and walking as well as tremor and dyskinesia scores.

Duration of the study for participants is approximately 4 to 5 days including 1-2 outpatient visits and a 3-day inpatient hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Have idiopathic Parkinson's disease treated with levodopa and experiencing motor fluctuations
* Response to levodopa had to be documented by a 10 percent increase in finger or foot tapping speed

Exclusion Criteria:

* Clinically significant cardiovascular, cerebrovascular, hepatic and renal diseases
* Psychosis
* Allergy to apomorphine or 5ht3 inhibitors
* Prolonged qt interval
* Pregnancy/breast-feeding
* Hemodynamic instability
* Severe nausea
* Alcohol/drug abuse
* Other unstable medical conditions

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Effects on parkinsonism measured with finger and foot tapping speed

CONTACTS AND LOCATIONS:
Overall Officials: John G. Nutt, MD, Principal Investigator — Professor of Neurology, Oregon Health and Science University; Steven Gunzler, MD, Principal Investigator — Fellow and Clinical Instructor in Neurology, Oregon Health and Science University
Locations (1):
- Department of Neurology, Oregon Health and Science University, Mail Code OP32, 3181 SW Sam Jackson Park Road, Portland, Oregon, United States

REFERENCES:
- [Derived] Gunzler SA, Koudelka C, Carlson NE, Pavel M, Nutt JG. Effect of low concentrations of apomorphine on parkinsonism in a randomized, placebo-controlled, crossover study. Arch Neurol. 2008 Feb;65(2):193-8. doi: 10.1001/archneurol.2007.58. PMID 18268187